CLINICAL TRIAL: NCT00161941
Title: Open-label Multicenter Phase 3B Follow-up Study to Investigate the Antibody Response to Hepatitis B, Acellular Pertussis Toxin and Inactivated Poliovirus Antigens One Month After the 4th Hexavac® Vaccination in Healthy Children, Who Participated in the NeisVac-C Non-interference Study 216
Brief Title: Follow-up Study on the Antibody Response to Hepatitis B, Acellular Pertussis Toxin and Inactivated Poliovirus Antigens 1 Month After the 4th Hexavac® Vaccination in Healthy Children, Who Participated in NeisVac-C Study 216
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Other Study IDs: 224
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Meningococcal Meninigitis, Serogroup C
Keywords: Meningococcal Vaccine; Meningococcal Meningitis, Serogroup C; Neisseria Meningitidis
MeSH Terms: conditions — Meningitis, Meningococcal

SUMMARY:
The primary aim of the study is to show that the antibody response to hepatitis B, acellular pertussis toxin and inactivated poliovirus antigens after the 4th vaccination with Hexavac® is not influenced by the concomitant administration of NeisVac-C.

ELIGIBILITY:
Inclusion Criteria:

Study subjects who completed study 216 will be eligible for participation in this study if:

* they received all 3 vaccinations with Hexavac during study 216 and the 4th Hexavac vaccination outside the study
* the subject's parent(s)/legal guardian(s) understands the study and has provided written informed consent for his/her child's study participation;
* a blood draw was performed after the 3rd vaccination during study 216.

Exclusion Criteria:

Study subjects will be excluded from participation in this study if:

* they have received any vaccination containing hepatitis B, poliovirus or acellular pertussis toxin antigens other than Hexavac
* they have received a blood transfusion or immunoglobulins during the period from 28 days prior to the 4th Hexavac vaccination until study entry
* they have received another vaccine during the period from 28 days prior to the 4th Hexavac vaccination until study entry
* they are concurrently participating in or have participated in a clinical trial with an investigational medicinal product since the completion of study 216
* they suffer from a disease (e.g. autoimmune disease) or were undergoing a form of treatment that may be expected to influence immunological functions since the completion of study 216
* they have received systemic corticosteroids during the period from 28 days prior to the 4th Hexavac vaccination until study entry.

Ages: 5 Months to 22 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 321
Dates: Start 2003-06; Study Completion 2003-12

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Behre, MD, Principal Investigator — Private practice, Hauptstrasse, Kehl, Germany
Locations (11):
- Grieskirchner Strasse 17, Wels, Austria
- Germany (10):
  - Neuschwansteinstrasse 5, Augsburg
  - Marktplatz 3, Bad Saulgau
  - Hauptrasse 9, Bietigheim-Bissingen
  - Rheinstrasse13, Ettenheim
  - Solothurner Strasse 2, Heilbronn
  - Hauptrasse 240, Kehl
  - Löpsinger Strasse 8, Nördlingen
  - Tuchbergstrass 2, Oberndorf / Neckar
  - Falkensteiner Str. 24, Roding
  - Berneckstrasse 19, Schrammberg